CLINICAL TRIAL: NCT02267720
Title: Survival Rate and Cost Effectiveness From Two Different Materials of GIC Using in Occlusol-proximal ART Restorations in Primary Molars
Brief Title: Occlusal-proximal ART Restorations in Primary Molars Using 2 Different Kinds of GIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Professor of Paediatric Dentistry, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USPARTOP2014
Record Dates: First submitted 2014-10-14; First posted 2014-10-17 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Dental Caries
Keywords: Dental Atraumatic Restorative Treatment; Glass ionomer cement; Occlusal-proximal leasons; Primary molars
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketac Molar (Active Comparator): Occlusal-proximal ART restorations - Ketac Molar
  Interventions: Procedure: Occlusal-proximal ART restorations - Vitro Molar
- Vitro Molar (Experimental): Occlusal-proximal ART restorations - Vitro Molar
  Interventions: Procedure: Occlusal-proximal ART restorations - Ketac Molar

INTERVENTIONS:
Procedure: Occlusal-proximal ART restorations - Ketac Molar — Occlusal-proximal ART restorations - Ketac Molar
  Arms: Vitro Molar
Procedure: Occlusal-proximal ART restorations - Vitro Molar — Occlusal-proximal ART restorations - Vitro Molar
  Arms: Ketac Molar

SUMMARY:
The aim of this research is to investigate the survival rate and cost effectiveness of two brands of GIC as occlusal-proximal ART restorations. Also the survival rate of the tooth will be investigated.

DETAILED DESCRIPTION:
Sampling procedure:

This study was approved by the research ethics committee of the School of Dentistry (University of São Paulo, Brazil) and a written informed consent will be obtained from the parents or legal guardians of the participating children. The sample size was calculated based on the minimum difference of 10% in the success rate between the control and treatment groups after 1 year of follow-up, with and α of 5% and power (strength) of 80% using paired test. According to the sample size calculation 150 children aged from 5-8 years old attending public schools from the city of Barueri in the state of São Paulo, Brazil will be selected.

To be included in this study the following criteria must be followed: healthy, cooperative children with at least one occlusal carious lesion in a primary molar extending to the dentin with dimensions not greater than 2 mm occluso-cervical and with an intact edge list. Also, to be included the tooth cannot present ulcer, abscess, fistula, or pathological mobility.

Implementation:

One occlusal restoration per child will be included in this study. If the selected children present more cavities, they will be referred to the health centre of the municipality of Barueri or will be treated by the operators of this research during the training week. All the occlusal and proximal-ART restorations will be performed by two operators on the school premisses3. The operators will be final year dental students who will be previously trained to perform ART and to mix the GIC according to the manufacturers' protocol. Additionally, a try-out week will be included to give the operators the opportunity to familiarise themselves with the local conditions prior to the start of the operative phase of the study. The operators will be assisted by a local dentist and a dentist assistant, who will be previously trained to mix the GIC according to the manufacturers' protocol. The children will be randomly assigned into three groups: Fuji IX, Maxxion R, and Vitro Molar and the GIC brand used in each child will be assigned by a random list. The operators are blind for the GIC brand.

Treatment procedure:

The ART technique will be performed according to the ART guidelines proposed by Frencken (2014)8. No local anaesthesia will be used during treatment. The plaque will be removed and an enamel hatchet will be used to make access to underlying softened dentine. Infected carious dentin will be removed with hand instruments. The use of hand instruments on the dentin surface results in a smear layer and need to be removed by the use of dentine conditioner. The liquid component of the hand-mixed powder-liquid GIC, containing the acid component, will be used and saliva isolation will be done with cotton wool rolls. The cavities will be restored with one of the three GIC brands: Fuji IX (GC Europe, Leuven, BE), Maxxion R (FGM, Rio de Janeiro, BR) and Vitro Molar (DHL, Rio de Janeiro, BR). The GICs will be hand mixed according to the manufacturers´ instructions (powder/liquid ratio 1:1) and will be inserted into the cavity with a conventional application instrument. A thin layer of petroleum jelly will be rubbed over the index finger and the restoration will be pressed for 20 seconds. The material will include sealing pits and the fissure. After preparing for a balanced occlusion, a new layer of petroleum jelly will be applied to the GIC restoration17. The amount of GIC used, element number, cavity dimension and dmft will be recorded. The duration of the restorative procedure will be recorded with a stop watch. The participating children will be instructed not to eat for one hour after the restoration is placed.

Estimation of cost-effectiveness:

Effectiveness will be measured in terms of the retention rate. This study will report only the preliminary results after 1 month, but the other follow-ups will be done every 6 months up to 3 years. The average cost per restoration will be estimated. Costs of equipment, autoclave and hand instruments, disposables (hand gloves, face masks, cotton wool rolls), articulating paper and petroleum jelly used for the restorations are equal for all the three GIC groups and will be excluded. There will be no labour costs for the operators. The material cost (powder-liquid GICs) will be estimated per restoration.

Evaluation:

The retention rate of the restorations will be evaluated after 1 month according to the modified version of Roeleveld et al. (2006) criteria (Table 1). A restoration will be considered as 'failure' when there is a defect in the filling, when secondary caries are observed, when the restoration is not present or when the pulp is inflamed. When the restoration is still present or a slight defect is observed, it will be considered as 'success'. When the tooth is unavailable for evaluation, it will be censored. All evaluations will be carried out by one independent evaluator, who did not restore the cavities, trained and calibrated by a benchmark.

The cost effectiveness will be evaluated. The total price of each GIC brand, used to insert into the cavities will be compared to the retention rate of the restorations9.

ELIGIBILITY:
Inclusion Criteria:

- the presence of at least one occluso-proximal carious lesion in a primary molar reaching dentin, but no larger than 2mm mesio-distal, 2.5mm bucco-lingual and occluso-cervical.

Exclusion Criteria:

* cases of pulp exposure, non-cooperative behaviour, pain, mobility, swelling, fistula or a lesion that cannot be cleaned with hand instruments, and absence of an adjacent tooth.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Survival rate of ART occluso-proximal restoration | Every 6 months up to 2 years
Survival rate of primary molar after ART restoration | Every 6 months up to exfoliation of the tooth
Cost effectiveness of two brands of GIC in occluso-proximal ART restorations | After 2 years

SECONDARY OUTCOMES:
Relation between approximal contact and survival rate | After 2 years
Relation between ICDAS adjacent tooth and survival rate | After 2 years
Relation between occlusal contact and survival rate | After 2 years
Difference between the two operators | After 2 years
Relation between contamination and survival rate | After 2 years
Relation between location of the teeth and survival rate | After 2 years
  Up or lower jaw, left or right side
Relation between the volume of the cavity after preparation and the survival rate | After 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, prof., Principal Investigator — University of Sao Paulo

REFERENCES:
- [Result] Bonifacio CC, Hesse D, Raggio DP, Bonecker M, van Loveren C, van Amerongen WE. The effect of GIC-brand on the survival rate of proximal-ART restorations. Int J Paediatr Dent. 2013 Jul;23(4):251-8. doi: 10.1111/j.1365-263X.2012.01259.x. Epub 2012 Aug 14. PMID 22891625
- [Result] Raggio DP, Hesse D, Lenzi TL, Guglielmi CA, Braga MM. Is Atraumatic restorative treatment an option for restoring occlusoproximal caries lesions in primary teeth? A systematic review and meta-analysis. Int J Paediatr Dent. 2013 Nov;23(6):435-43. doi: 10.1111/ipd.12013. Epub 2012 Nov 28. PMID 23190278